CLINICAL TRIAL: NCT04796090
Title: Genital Warts is Related With Sexual Dysfunction and Sexual Distress in Adolescence
Brief Title: Genital Wart and Sexuality in Adolescence
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Esin Merve Erol Koç, Principal Investigator, Ankara City Hospital Bilkent
Other Study IDs: E1-20-1000
Record Dates: First submitted 2021-03-10; First posted 2021-03-12 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Adolescent Development; Genital Wart; Sexual Dysfunction; Sexual Disorder, Physiological
Keywords: Genital wart; Female sexual dysfunction; Late adolescence; Sexuality related distress
MeSH Terms: conditions — Condylomata Acuminata; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adolescents with genital warts (Study Group): The Study group included adolescents who was diagnosed as positive for genital warts during the examination.
  Interventions: Other: Clinical assessment
- Healthy adolescents (Control Group): The Control group was composed of healthy adolescents who admitted for only contraceptive counselling.
  Interventions: Other: Clinical assessment

INTERVENTIONS:
Other: Clinical assessment — FSFI, ASEX and FSDS scores were compared between the adolescents with (Study group) or without (Control group) genital warts.

SUMMARY:
The adolescence is a landmark in perceiving the sexuality and awareness about the sexual experiences. Genitals warts were shown to be a potential risk to impair the sexual functions in women. Adolescence is a vulnerable period in which the individuals may be prone to the negative effects of the disorders affecting sexual functions such as genital warts. The current study aimed to investigate the impact of genital warts on sexual functions in female adolescents.

DETAILED DESCRIPTION:
This current study aimed to elucidate the impact of genital warts on female sexual function in adolescence. The current study also targeted to reveal whether there is any correlation between the genital warts and the female sexual dysfunction, as well as the sexuality related distress. The current study is conducted at Youth Center Outpatient Clinic of Ankara City Hospital which is a high-volume tertiary health care center in Turkey. The study was prospectively designed and data were collected between the 1 August 2020 and 1 February 2021. Totally 90 female adolescents between the age of 17-21 who had regular sexual intercourse with heterosexual partners were included. The Study group composed of 45 adolescents who had genital warts and the Control group included 45 healthy adolescents. Female sexual function Index (FSFI), Arizona Sexual Experiences Scale (ASEX) and Female Sexual Dysfunction Scale (FSDS) scores were compared between the two groups to evaluate the sexual functions. Difference between two independent means (two groups) power analysis demonstrated that this study achieved a power of 0.99, 0.98 , 0.99 with a 5% level of significance for comparison of 45 adolescents with genital warts and 45 healthy adolescents in terms of FSFI, ASEX, and FSDS scores, respectively.

ELIGIBILITY:
Inclusion Criteria:

* The Study group included adolescents who was diagnosed as positive for genital warts during the examination.
* The Control group was composed of healthy adolescents who admitted for contraceptive counselling.

Exclusion Criteria:

* Chronical disease including rheumatological diseases, renal failure, diabetes mellitus, hypertension, dyslipidemia, obesity, thyroid dysfunction, cardiopulmonary diseases, malignancy, cerebrovascular diseases, psychiatric and mental disorders, cerebrovascular diseases, inflammatory bowel diseases.
* Drug administration which may interfere sexual function.
* Surgical intervention to genital organs.
* History of pregnancy, delivery, and/or breastfeeding.

Ages: 17 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — The study is aimed to elucidate female adolescents' sexual functions.
Study Population: The current study included 45 adolescents with the diagnosis of genital warts as the Study group and 45 healthy adolescents as the Control group.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Female Sexual Function Index | Through study completion, an average of 6 months
  Questionnaire score with minimum and maximum levels of 2.4 and 36 points,respectively. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Arizona Sexual Experiences Scale | Through study completion, an average of 6 months
  Questionnaire score with minimum and maximum levels of 5 and 30 points,respectively. Higher scores mean a worse outcome.
Female Sexual Distress Scale-Revised | Through study completion, an average of 6 months
  Questionnaire score with minimum and maximum levels of 0 and 50 points,respectively. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Esin Merve Erol Koç, MD, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data belonging to participants only will be available to any researcher or editorial review board if needed.

REFERENCES:
- [Result] Graziottin A, Serafini A. HPV infection in women: psychosexual impact of genital warts and intraepithelial lesions. J Sex Med. 2009 Mar;6(3):633-45. doi: 10.1111/j.1743-6109.2008.01151.x. Epub 2009 Jan 13. PMID 19170869
- [Result] McCabe MP, Sharlip ID, Atalla E, Balon R, Fisher AD, Laumann E, Lee SW, Lewis R, Segraves RT. Definitions of Sexual Dysfunctions in Women and Men: A Consensus Statement From the Fourth International Consultation on Sexual Medicine 2015. J Sex Med. 2016 Feb;13(2):135-43. doi: 10.1016/j.jsxm.2015.12.019. PMID 26953828
- [Result] McGahuey CA, Gelenberg AJ, Laukes CA, Moreno FA, Delgado PL, McKnight KM, Manber R. The Arizona Sexual Experience Scale (ASEX): reliability and validity. J Sex Marital Ther. 2000 Jan-Mar;26(1):25-40. doi: 10.1080/009262300278623. PMID 10693114
- [Result] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Result] Greydanus DE, Matytsina L. Female sexual dysfunction and adolescents. Curr Opin Obstet Gynecol. 2010 Oct;22(5):375-80. doi: 10.1097/GCO.0b013e32833d9418. PMID 20706119
- [Result] Derogatis L, Clayton A, Lewis-D'Agostino D, Wunderlich G, Fu Y. Validation of the female sexual distress scale-revised for assessing distress in women with hypoactive sexual desire disorder. J Sex Med. 2008 Feb;5(2):357-64. doi: 10.1111/j.1743-6109.2007.00672.x. Epub 2007 Nov 27. PMID 18042215
- [Result] O'Sullivan LF, Byers ES, Brotto LA, Majerovich JA, Fletcher J. A Longitudinal Study of Problems in Sexual Functioning and Related Sexual Distress Among Middle to Late Adolescents. J Adolesc Health. 2016 Sep;59(3):318-324. doi: 10.1016/j.jadohealth.2016.05.001. Epub 2016 Jun 16. PMID 27320034